CLINICAL TRIAL: NCT01859065
Title: "Anticipatory Guidance in the Nursery and Its Impact on Non-urgent Emergency Department Visits"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx-Lebanon Hospital Center Health Care System (Other)
Responsible Party: Principal Investigator, Kelly Kamimura-Nishimura, MD, Pediatric Resident, Bronx-Lebanon Hospital Center Health Care System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 09 15 11 10
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Health Knowledge, Attitudes, Practice; Sneezing; Constipation; Nasal Congestion and Inflammations
Keywords: Non-urgent ED visits; Neonates; Newborn care
MeSH Terms: conditions — Behavior; Sneezing; Constipation; Nasal Obstruction; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Mothers receive routine anticipatory guidance
  Interventions: Behavioral: Routine
- Intervention (Experimental): Mothers receive video-based and handout-based anticipatory guidance regarding non-urgent problems in addition to the routine anticipatory guidance
  Interventions: Behavioral: Intensified anticipatory guidance

INTERVENTIONS:
Behavioral: Intensified anticipatory guidance — Mothers receive video-based and handout-based anticipatory guidance regarding non-urgent problems in addition to the routine anticipatory guidance
  Arms: Intervention
Behavioral: Routine — Routine anticipatory guidance (control)
  Arms: Control

SUMMARY:
Kennedy et al, in a study of pediatric Emergency Department (ED) use by newborns less than 14 days of age, revealed that half of all visits in this population were non-acute problems. Other pediatric ED utilization studies have shown similar findings in that 32% to 72% of all visits were for non-urgent problems.

Many studies have found that primiparity and young maternal age are associated with non-acute ED presentations. A recent factor that has been investigated is the effect of early neonatal discharge. Some other factors are nonwhite mothers and mothers on Medicaid. Zandieh et al, found additional predisposing determinants for non-urgent ED visits, such as single parenthood, Hispanic ethnicity, and having perceptions that their child's overall physical health was poor.

Paradis et al found that parents receiving a video intervention rated higher confidence with specific infant care skills and reported feeling better prepared to care for their baby, compared to parents receiving only handouts. However, there isn't any reported study that evaluates the benefits of receiving both, a video intervention along with handouts.

Aim: to demonstrate whether conducting anticipatory guidance related to non-urgent problems will reduce non-urgent ED visits, compared to care as usual (CAU) anticipatory guidance (Sudden Infant Death Syndrome and Shaken Baby Syndrome videos; and unstructured talk about jaundice, vaccinations, appointments, care of umbilical stump, normal urination and bowel movement, fever).

DETAILED DESCRIPTION:
Inclusion Criteria: Mother of a newborn in the Well Baby Nursery (WBN) of Bronx-Lebanon Hospital Center during the 4-month recruitment period of the study.

Exclusion Criteria:

1. Mothers selected for video-based anticipatory guidance that have a hearing/vision impairment.
2. Mothers selected for handout-based anticipatory guidance who speak a language other than Spanish or English.

Primary outcome measure: reduction in non-urgent ED visits in mothers who received the intervention (video-based and handout-based anticipatory guidance regarding non-urgent problems), compared to the control group (received CAU anticipatory guidance)

Secondary outcome measure: improvement in parental knowledge, attitude and behaviors related to non-urgent problems as a result of receiving anticipatory guidance (video and handouts) regarding non-urgent problems;

ELIGIBILITY:
Inclusion Criteria:

* Mother of a newborn in the WBN of Bronx-Lebanon Hospital Center during the 4-month recruitment period of the study

Exclusion Criteria:

* Mothers selected for video-based anticipatory guidance that have a hearing/vision impairment.
* Mothers selected for handout-based anticipatory guidance who speak a language other than Spanish or English.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Non-urgent ED visits by neonates | 1 month
  Reduction in non-urgent ED visits in mothers who received the intervention (video-based and handout-based anticipatory guidance regarding non-urgent problems), compared to the control group (received CAU anticipatory guidance)

SECONDARY OUTCOMES:
Changes in caregivers' knowledge and attitude | 1 month
  Improvement in parental knowledge, attitude and behaviors related to non-urgent problems as a result of receiving anticipatory guidance (video and handouts) regarding non-urgent problems

CONTACTS AND LOCATIONS:
Overall Officials: Ayoade Adeniyi, MD, Principal Investigator — Bronx-Lebanon Hospital Center
Locations (1):
- Bronx Lebanon Hospital Center, The Bronx, New York, United States

REFERENCES:
- [Background] Paradis HA, Conn KM, Gewirtz JR, Halterman JS. Innovative delivery of newborn anticipatory guidance: a randomized, controlled trial incorporating media-based learning into primary care. Acad Pediatr. 2011 Jan-Feb;11(1):27-33. doi: 10.1016/j.acap.2010.12.005. PMID 21272821
- [Background] Rosenthal MS, Lannon CM, Stuart JM, Brown L, Miller WC, Margolis PA. A randomized trial of practice-based education to improve delivery systems for anticipatory guidance. Arch Pediatr Adolesc Med. 2005 May;159(5):456-63. doi: 10.1001/archpedi.159.5.456. PMID 15867120
- [Background] Schuster MA, Duan N, Regalado M, Klein DJ. Anticipatory guidance: what information do parents receive? What information do they want? Arch Pediatr Adolesc Med. 2000 Dec;154(12):1191-8. doi: 10.1001/archpedi.154.12.1191. PMID 11115301
- [Background] Barkin SL, Scheindlin B, Brown C, Ip E, Finch S, Wasserman RC. Anticipatory guidance topics: are more better? Ambul Pediatr. 2005 Nov-Dec;5(6):372-6. doi: 10.1367/A04-2131R1.1. PMID 16302840
- [Background] Kennedy TJ, Purcell LK, LeBlanc JC, Jangaard KA. Emergency department use by infants less than 14 days of age. Pediatr Emerg Care. 2004 Jul;20(7):437-42. doi: 10.1097/01.pec.0000132216.65600.1b. PMID 15232243
- [Background] Pomerantz WJ, Schubert CJ, Atherton HD, Kotagal UR. Characteristics of nonurgent emergency department use in the first 3 months of life. Pediatr Emerg Care. 2002 Dec;18(6):403-8. doi: 10.1097/00006565-200212000-00001. PMID 12488831
- [Background] Zandieh SO, Gershel JC, Briggs WM, Mancuso CA, Kuder JM. Revisiting predictors of parental health care-seeking behaviors for nonurgent conditions at one inner-city hospital. Pediatr Emerg Care. 2009 Apr;25(4):238-243. doi: 10.1097/pec.0b013e31819e350e. PMID 19382324
- [Background] Rudominer A. Reducing Newborn Office Visits and Improving Satisfaction through Parent Education and Learning Communities. Perm J. 2009 Summer;13(3):25-30. doi: 10.7812/TPP/08-096. No abstract available. PMID 20740085
- [Derived] Kamimura-Nishimura K, Chaudhary V, Olaosebikan F, Azizi M, Galiveeti S, Adeniyi A, Neugebauer R, Hagmann SH. Does Nursery-Based Intensified Anticipatory Guidance Reduce Emergency Department Use for Nonurgent Conditions in the First Month of Life? A Randomized Controlled Trial. Int J Pediatr. 2016;2016:8356582. doi: 10.1155/2016/8356582. Epub 2016 Apr 24. PMID 27212955